CLINICAL TRIAL: NCT03391531
Title: Placebo-controlled, Randomized, Double-blind Trial of Transversus Abdominis Plane Block on Pain After Laparoscopic Cholecystectomy
Brief Title: Analgesic Effect of TAP Block After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of the department of Anesthesiology, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAPLAPCHOL
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Analgesia
Keywords: surgery: laparoscopic cholecystectomy; analgesia: postoperative; locoregional analgesia: transversus abdominis plane block; opioid: side effects

STUDY DESIGN:
Intervention Model Description: two groups : treatment group (TAP block with local anesthestic) compared to control group (TAP block with saline)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Person who prepares the study solution is involved neither in any step of the care of the patient neither in the collection of the study parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levobupivacaine (Active Comparator): Echo-guided bilateral subcostalTAP block will be performed using levobupivacaine [Chirocaine®] 0.375% Epi 1/200000.
  Interventions: Procedure: Bilateral subcostal TAP block
- Saline (Placebo Comparator): Echo-guided bilateral subcostal TAP block will be performed with saline Epi 1/200000 in the control group.
  Interventions: Procedure: Bilateral subcostal TAP block

INTERVENTIONS:
Procedure: Bilateral subcostal TAP block — Echo-guided infiltration of a local anesthetic solution in the plane located between the transversus abdominis muscle and the rectus abdominis muscle

SUMMARY:
TAP block is a locoregional analgesic technique that consists of infiltrating a local anesthetic solution between the muscle layers of the abdominal wall. This block produces prolonged parietal analgesia.

The aim of the study is to evaluate whether infiltration of the abdominal wall using TAP block reduces postoperative pain and postoperative analgesic consumption, and improves patient comfort after laparoscopic cholecystectomy. This effect will be clinically relevant only if parietal pain predominates postoperatively.

DETAILED DESCRIPTION:
Between 10 and 20% of the Western population suffer from gallstones. When a surgical operation (cholecystectomy) is necessary, the removal of the gallbladder is done by laparoscopy in 95% of cases. The risk of having to undergo this operation increases with age and on average women are twice as likely as men to have to undergo surgery. In Belgium, only 4% of these laparoscopic cholecystectomies are performed as one day hospitalization. Although this operation is considered a minor surgery, patients sometimes report intense postoperative pain that may encourage them to spend a night in the hospital. Better management of postoperative pain could increase the number of outpatient procedures. A large individual variability in pain intensity is observed after this surgical procedure. Three types of pain can be associated with this surgery: parietal pain secondary to the incisions of the wall necessary for the introduction of the surgical instruments; deep visceral pain, difficult to localize and secondary to surgical trauma in the area of dissection of the gall bladder; and scapular pain, a projected pain secondary to the irritation of the diaphragm by CO2-pneumoperitoneum. The temporal characteristics and intensity of these three types of pain are different. Some report a predominance of parietal pain, while for others visceral pain is most intense.

The Transversus Abdominis Plane (TAP) block is a loco-regional analgesia technique that consists of infiltrating a local anesthetic solution between the plane of the transversus abdominis muscle and the internal oblicus muscle, laterally at the level of the triangle of Petit. The sensory nerves of the abdominal wall pass through this plane. This technique produces long-lasting analgesia, between 24-36 hours. Only the nerves responsible for the innervation of the abdominal wall are blocked by this infiltration. The metameric extension of parietal analgesia varies from one study to another, especially depending on the site of infiltration. After posterior TAP block, parietal analgesia concerns the infra-umbilical abdominal wall, but can reach in some cases the dermatome T-8. When the surgery involves the supra-umbilical abdominal wall, the TAP block is performed at the subcostal level to block the nerve branches T-6 to T-10. Infiltration is then performed between the transverse muscle and the rectus abdominis at the lateral end of this muscle.

Several studies have evaluated the efficacy of TAP block for analgesia after laparoscopic cholecystectomy. Controversial results have been reported. These controversies can be explained in part by the type of TAP block used: lateral versus subcostal approach which appears more appropriate for laparoscopic cholecystectomy (supra-umbilical parietal incisions). In addition, effective multimodal analgesia, a recommended good medical practice, is not always used in these studies. This strategy, by effectively reducing postoperative pain, may make the clinical utility of TAP block irrelevant. Finally, in case of predominance of parietal pain on visceral pain, the clinical relevance of the TAP block should be objectified. In the opposite case (predominance of visceral pain), TAP block would be much less effective.

2.2 Purpose of the study. The purpose of this study is to evaluate the analgesic efficacy of TAP subcostal block after laparoscopic cholecystectomy. The effectiveness of the TAP block will confirm the importance of the parietal pain component after this type of surgery. Decreases in postoperative pain and postoperative opioid consumption, possibly associated with a decrease in morphine side effects (nausea, vomiting, sedation, fatigue), may be conducive to the development of outpatient laparoscopic cholecystectomy.

2.3 General description. This randomized double-blind placebo-controlled study will include two groups of 20 patients: the TAP block will be performed in a group using a local anesthetic solution (levobupivacaine [Chirocaine®] 0.375% Adr 1/200000) in the " treatment " group and with saline Adr 1/200000 in the control group.

ELIGIBILITY:
Inclusion Criteria:

- all patients aged 18-75 yo scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Coagulation disorders
* Refusal of participation expressed by the patient
* Fibromyalgia
* Preoperative morphine treatment
* Contraindications to local anesthetics: epilepsy, severe cardiac conduction block (2nd and 3rd degree AVB ), allergy
* Contraindications to NSAIDs: renal failure, allergy, ischemic heart disease, stroke

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative opioid consumption | 24 hours
  opioid given as an IV titration in the PACU, and opioid po on the ward

SECONDARY OUTCOMES:
postoperative pain intensity | 24 hours
  postoperative pain will be separated out in parietal, visceral, and shouldertip pain; pain will be measured on 0-10 visual analog scale
postoperative nausea and vomiting | 24 hours
  PONV measured on 0-10 visual analog scale
postoperative fatigue | 24 hours
  measured on 0-10 visual analog scale
intraoperative sevoflurane consumption | 2 hours
  end-tidal sevoflurane concentration will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Joris, M.D., Principal Investigator — Department of Anesthesiology, CHU Liege, Belgium
Locations (1):
- CHU Liege,, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No